CLINICAL TRIAL: NCT02402062
Title: A Phase II Study to Assess the Activity and Safety of TH-302 in Combination With Sunitinib in Treatment-naïve Patients With Well- and Moderately-differentiated Metastatic Pancreatic Neuroendocrine Tumours (pNET)
Brief Title: A Study to Assess the Safety and the Efficacy of the Combination of TH-302 and Sunitinib in Neuroendocrine Pancreatic Tumours
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Grupo Espanol de Tumores Neuroendocrinos (Other)
Collaborators: Threshold Pharmaceuticals (Industry); Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GETNE-1408; 2014-004072-30 (EudraCT Number)
Record Dates: First submitted 2015-02-26; First posted 2015-03-30 (Estimated); Results first posted 2020-07-27 (Actual); Last update posted 2020-07-27 (Actual); Status verified 2020-07

CONDITIONS: Neuroendocrine Tumors; Pancreatic Neoplasms
Keywords: pNET
MeSH Terms: conditions — Neuroendocrine Tumors; Pancreatic Neoplasms; Neuroectodermal Tumors, Primitive | interventions — TH 302; Sunitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- TH-302 + Sunitinib (Experimental): TH-302 + Sunitinib. Single arm Study.
  Interventions: Drug: TH-302 + Sunitinib

INTERVENTIONS:
Drug: TH-302 + Sunitinib — Combination of the two drugs in cycles of 28 days, described as follows:
  Sunitinib: 37,5 mg/day Oral everyday of each 28 day cycle.
  TH-302: 340 mg/m2 IV on days 8, 15 and 22 of each cycle.
  Other Names: TH-302 + Sutent

SUMMARY:
The purpose of this study is to determine the safety and the efficacy of the combination of the drugs TH-302 and sunitinib in metastatic neuroendocrine tumours.

DETAILED DESCRIPTION:
The purpose of this study is to determine the safety and the efficacy of the combination of the drugs TH-302 and sunitinib in Treatment-naïve patients with well- and moderately-differentiated metastatic Pancreatic Neuroendocrine Tumours (pNET).

ELIGIBILITY:
Inclusion Criteria:

* Male or female, 18 years of age or older.
* Eastern Cooperative Oncology Group (ECOG) performance status 0-1.
* Histologically proven diagnosis of pancreatic neuroendocrine tumors (pNET) with Ki67 assessment of ≤ 20% (well and moderately differentiated)
* Evidence of unresectable disease or metastatic disease. Locally advanced disease must not be amendable to resection or radiation therapy with curative intent.
* Patients may be treated with somatostatin analogues prior or during the trial. Concomitant or prior interferon treatment is not permitted.
* Documented progression disease by CT scan, magnetic resonance (MR) or Octreoscan in 12 months prior basal visit.
* Measurable disease as per RECIST. Measurable lesions that have been previously radiated will not be considered target lesions unless increase in size has been observed following completion of radiation therapy.
* Patient has to be able to swallow the medication.
* Life expectancy greater than 12 weeks.
* The definitions of minimum adequacy for organ function required prior to study entry are as follows:

  * Serum aspartate transaminase (AST) and serum alanine transaminase (ALT) ≤ 2.5 x upper limit of normal (ULN), or AST and ALT ≤ 5 x ULN if liver function abnormalities are due to underlying malignancy
  * Total serum bilirubin ≤ 1.5 x ULN
  * Serum albumin ≥ 3.0 g/dL
  * Absolute neutrophil count (ANC) ≥ 1500/µL
  * Platelets ≥ 100,000/µL
  * Hemoglobin ≥ 5,6 mmol/L (9.0 g/dL)
  * Creatinin clearance > 40 mL/min (Cockcroft and Gault formula)
* Adequate cardiac function: 12-lead ECG without pathologic findings (clinically significant alterations are allowed) and Echocardiogram / Normal multiple gated acquisition scan (MUGA) (LVEF> 50%)
* Signed and dated informed consent document indicating that the patient (or legally acceptable representative) has been informed of all the pertinent aspects of the trial prior to enrollment.
* Willingness and ability to comply with scheduled visits, treatment plans, laboratory tests, and other study procedures.

Exclusion Criteria:

* Previous treatments with chemotherapy, monoclonal antibodies anti-vascular endothelial growth factor (VEGF), tyrosine kinase inhibitors, mammalian target of rapamycin (mTOR) inhibitors, or interferon are not permitted for the advanced disease.
* Prior treatment on another hypoxia-activated prodrug under clinical trial.
* Major surgery, radiation therapy, or systemic therapy within 3 weeks of study randomization except palliative radiotherapy to non-target metastatic lesions.
* Prior high-dose chemotherapy requiring hematopoietic stem cell rescue.
* Immunosuppressive drugs such as cyclosporine, tacrolimus, azathioprine, or long-term oral glucocorticoids taken concurrently or within last 3 months prior to randomization
* Treatment with known inhibitors or inductors of cytochrome P450 3A4 (CYP3A4) or that prolong the QT interval in the previous 7 days.
* Prior radiation therapy to > 25% of the bone marrow.
* Current treatment on another clinical trial.
* Uncontrolled brain metastases, spinal cord compression, carcinomatous meningitis, or leptomeningeal disease. Patients should have completed surgery or radiation therapy for existing brain metastases, should not have documented increase in size over the previous 3 months prior to first dose of treatment on study and should be asymptomatic.
* Diagnosis of any second malignancy within the last 3 years, except for adequately treated basal cell or squamous cell skin cancer, or carcinoma in situ of the cervix.
* Any of the following within the 12 months prior to starting study treatment:

  * myocardial infarction,
  * severe/unstable angina,
  * coronary/peripheral artery bypass graft,
  * congestive heart failure class III or IV of the New York Heart Association (NYHA) or patients with clinical history of congestive heart failure class III or IV of the NYHA, unless an echocardiogram or MUGA in the previous 3 months to selection shows a LVEF ? 45 %
  * significant heart valve disease
  * cerebrovascular accident including transient ischemic attack
  * pulmonary embolus.
* Ongoing cardiac dysrhythmias of NCI Common Toxicity Criteria for Adverse Effects (CTCAE) grade ≥ 2, atrial fibrillation of any grade, or corrected QT interval (QTc) interval >450 msec for males or >470 msec for females.
* Hypertension that cannot be controlled by medications (>150/100 mmHg despite optimal medical therapy)
* Chronic obstructive pulmonary disease (COPD) or any other disease concurrent with hypoxemia or oxygen saturation < 90% after a march of two minutes.
* Current treatment with therapeutic doses of Coumadin (low dose Coumadin up to 2 mg PO daily for deep vein thrombosis prophylaxis is allowed).
* Known human immunodeficiency virus infection.
* Pregnancy or breastfeeding. All female patients with reproductive potential must have a negative pregnancy test (serum or urine) prior to inclusion.
* Previous allergic reaction to components structurally similar to TH-302 or sunitinib or any of the excipients of drugs.
* Non-healing wound, fistulae, active peptic ulcer or bone fracture.
* Other severe acute or chronic medical or psychiatric condition, or laboratory abnormality that would impart, in the judgment of the investigator, excess risk associated with study participation or study drug administration, or which, in the judgment of the investigator, would make the patient inappropriate for entry into this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2015-05-11 (Actual); Primary Completion 2018-05-31 (Actual); Study Completion 2020-01-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Enrique Grande, MD, Study Chair — Grupo Espanol de Tumores Neuroendocrinos
Locations (10):
- Spain (10):
  - Institut Catalá d'Oncologia L'Hospitalet, L'Hospitalet de Llobregat, Barcelona
  - Hospital Universitario Marqués de Valdecilla, Santander, Cantabria
  - Hospital Provincial de Castellón, Castellon, Valencia
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Hospital Universitario Virgen de las Nieves, Granada
  - Hospital Universitario Ramón y Cajal, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario La Paz, Madrid
  - Hospital Universitario Virgen de la Victoria, Málaga
  - Hospital Universitario Virgen del Rocío, Seville

REFERENCES:
- [Derived] Grande E, Rodriguez-Antona C, Lopez C, Alonso-Gordoa T, Benavent M, Capdevila J, Teule A, Custodio A, Sevilla I, Hernando J, Gajate P, Molina-Cerrillo J, Diez JJ, Santos M, Lanillos J, Garcia-Carbonero R. Sunitinib and Evofosfamide (TH-302) in Systemic Treatment-Naive Patients with Grade 1/2 Metastatic Pancreatic Neuroendocrine Tumors: The GETNE-1408 Trial. Oncologist. 2021 Nov;26(11):941-949. doi: 10.1002/onco.13885. Epub 2021 Jul 14. PMID 34190375

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Meeting eligibility criteria: 17 patients that meet the eligibility criteria were finally included
Groups:
- TH-302 + Sunitinib: TH-302 + Sunitinib. Single arm Study.
  TH-302 + Sunitinib: Combination of the two drugs in cycles of 28 days, described as follows:
  Sunitinib: 37,5 mg/day Oral everyday of each 28 day cycle.
  TH-302: 340 mg/m2 IV on days 8, 15 and 22 of each cycle.
Period: Overall Study
Arm/Group | TH-302 + Sunitinib
Started | 17
Completed | 17
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | TH-302 + Sunitinib
Number analyzed (Participants) | 17
Age, Continuous [Median (Standard Deviation); unit: Years] | 60.78 (10.78)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 11
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 17
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Spain | 17
ECOG PS [Count of Participants; unit: Participants] — The ECOG Performance Status is a simple measure of functional status. It has scores ranging from 0 to 5:
  0: Fully active, without restriction
  1. Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature
  2. Ambulatory and capable of all selfcare but unable to carry out any work activities; up and about more than 50% of waking hours
  3. Capable of only limited selfcare; confined to bed or chair more than 50% of waking hours
  4. Completely disabled; cannot carry on any selfcare; totally confined to bed or chair
  5. Death
  Participants
    grade 0 | 11
    grade 1 | 6
Electrocardiogram (ECG) [Count of Participants; unit: Participants] — QT interval longer than 450ms
  Participants | 17
Left ventricular ejection fraction (LVEF) [Count of Participants; unit: Participants] — Left ventricular ejection fraction (LVEF) higher than 50%
  Participants | 17
Abbreviated Charlson comorbidity index [Count of Participants; unit: Participants] — The Charlson comorbidity index predicts the one-year mortality for a patient who may have a range of comorbid conditions. Each comorbidity category has an associated weight (from 1 to 6), based on the adjusted risk of mortality or resource use, and the sum of all the weights results in a single comorbidity score for a patient. A score of zero indicates that no comorbidities were found. The higher the score, the more likely the predicted outcome will result in mortality or higher resource use. The total scores range from 0 to 37.
  Participants
    index 2 | 11
    index 3 | 4
    index 4 | 2
Peripheral arterial disease [Count of Participants; unit: Participants]
  Yes | 1
  No | 16
Diabetes [Count of Participants; unit: Participants]
  Yes | 5
  No | 12
Tumor histological grade [Count of Participants; unit: Participants] — grade I: cancer cells that resemble normal cells and aren't growing rapidly grade II: cancer cells that don't look like normal cells and are growing faster than normal cells grade III: cancer cells that look abnormal and may grow or spread more aggressively
  Participants
    Grade I | 2
    Grade II | 15
Ki-67 index [Count of Participants; unit: Participants] — KI-67 is a measure of the rate of tumor growth, the higher the rate of Ki-67 proliferation, the faster cells are dividing, and is another prognostic factor.
  Participants
    >10% | 8
    >2%-5% | 5
    >5%-10% | 4
Mitosis 10 HPF [Count of Participants; unit: Participants] — The mitotic index is the number of cells undergoing mitosis divided by the total number of cells noted per 10 high power fields.
  Participants
    Unknown | 6
    <2 | 6
    2-20 | 5
Primary tumor surgery [Count of Participants; unit: Participants]
  Yes | 6
  No | 11
Tumor stage at diagnosis [Count of Participants; unit: Participants] — stage 0: indicates that the cancer is where it started (in situ) and hasn't spread stage I: the cancer is small and hasn't spread anywhere else stage II: the cancer has grown, but hasn't spread stage III: the cancer is larger and may have spread to the surrounding tissues and/or the lymph nodes (part of the lymphatic system) stage IV: the cancer has spread from where it started to at least one other body organ; also known as "secondary" or "metastatic" cancer
  Participants
    II | 3
    III | 1
    IV | 13
Tumor relapse location [Count of Participants; unit: Participants]
  Hepatic | 12
  Extra-hepatic | 1
  Unknown | 4
Somatostanine analogues prior the trial [Count of Participants; unit: Participants]
  Yes | 7
  No | 10
Baseline concomitant medication [Count of Participants; unit: Participants]
  Yes | 16
  No | 1
Weight [Mean (Standard Deviation); unit: Kg] | 70.97 (15.01)
Height [Mean (Standard Deviation); unit: cm] | 166.71 (7.74)
Body mass index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 25.46 (4.75)
Body surface area (BSA) [Mean (Standard Deviation); unit: m^2] | 1.79 (0.2)
Blood pressure systolic (BPs) [Mean (Standard Deviation); unit: mm Hg] | 134.82 (10.95)
Blood pressure diastolic (BPd) [Mean (Standard Deviation); unit: mm Hg] | 79.12 (7.42)
Haemoglobin [Mean (Standard Deviation); unit: g/dL] | 13.82 (1.21)
White blood cells [Mean (Standard Deviation); unit: x10^9 cells/L] | 6.22 (2.17)
Absolute neutrophil count [Mean (Standard Deviation); unit: x10^9 cells/L] | 4.52 (1.84)
Absolute Lymphocytes count [Mean (Standard Deviation); unit: x10^9 cells/L] | 1.69 (0.41)
Platelet count [Mean (Standard Deviation); unit: x10^9 cells/L] | 202.94 (77.34)
Sodium blood levels [Mean (Standard Deviation); unit: mmol/L] | 139.22 (3.06)
Potassium blood levels [Mean (Standard Deviation); unit: mmol/L] | 4.35 (0.35)
Calcium blood levels [Mean (Standard Deviation); unit: mmol/L] | 9.18 (1.83)
Magnesium blood levels [Mean (Standard Deviation); unit: mmol/L] | 1.9 (0.38)
Glucose [Mean (Standard Deviation); unit: mmol/L] | 133.44 (59.92)
Creatinine [Mean (Standard Deviation); unit: mg/dL] | 0.76 (0.17)
Aspartate AST (SGOT) [Mean (Standard Deviation); unit: u/L] | 48.95 (40.18)
Alanine transaminase ALT (SGPT) [Mean (Standard Deviation); unit: u/L] | 69.63 (61.12)
AST (SGOT)/ ALT (SGPT) (baseline) [Mean (Standard Deviation); unit: Ratio (arbitrary units)] | 0.83 (0.30)
Total bilirubin [Mean (Standard Deviation); unit: mg/dL] | 0.86 (0.58)
Gamma-glutamyltransferase (GGT) [Mean (Standard Deviation); unit: u/L] | 351.25 (488.76)
Alkaline phosphatase (AP) [Mean (Standard Deviation); unit: u/L] | 201.64 (183.95)
Albumin [Mean (Standard Deviation); unit: mg/dL] | 4.28 (0.43)
Lactate dehydrogenase (LDH) [Mean (Standard Deviation); unit: u/L] | 216.88 (83.41)
CG a tumor marker [Mean (Standard Deviation); unit: ng/L] | 474.41 (626.35)
Enolase 1 [Mean (Standard Deviation); unit: ng/mL] | 31.92 (31.08)
Time between diagnosis (anatomical pathology) and treatment initiation in months [Mean (Standard Deviation); unit: months] | 14.12 (22.72)
Time between diagnosis (anatomical pathology) and surgery in months [Mean (Standard Deviation); unit: months] | 1.1 (2.94)
Time between diagnosis (anatomical pathology) and CT relapse in months [Mean (Standard Deviation); unit: months] | 8.9 (13.77)

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate
Description: Objective response rate: percentage of patients in whom a complete response (CR) or a partial response (PR) is confirmed according Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 criteria in relation to the total of the analyzed population.
  Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions
Time Frame: approximately 36 months
Measure: Count of Participants; unit: Participants
Arm/Group | TH-302 + Sunitinib
Number analyzed (Participants) | 17
Participants
  CR or PR | 3
  SD or PD | 14

2. Secondary Outcome: Progression Free Survival (PFS)
Description: Time between the start of study treatment to date of the first objective evidence of radiological progression or patient death due to any cause; which comes first.
Time Frame: approximately 36 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | TH-302 + Sunitinib
Number analyzed (Participants) | 17
months | 10.38 [2.66 to 18.1]

3. Secondary Outcome: Time to Tumour Progression (TTP)
Description: It is defined as the time between the start of study treatment to date of the first objective evidence of radiological progression.
Time Frame: approximately 36 months
Measure: Median (Full Range); unit: months
Arm/Group | TH-302 + Sunitinib
Number analyzed (Participants) | 17
months | 5.32 [1.69 to 13.55]

4. Secondary Outcome: Duration of Response (DR)
Description: It is defined as the time between the start from the first documentation of objective response (CR or PR) which is subsequently confirmed until the first objective evidence of radiological progression or death from any cause. DR is calculated only in the subgroup of patients with an objective response (CR + PR).
Time Frame: approximately 36 months
Measure: Median (Full Range); unit: months
Arm/Group | TH-302 + Sunitinib
Number analyzed (Participants) | 3
months | 18.48 [4.20 to 38.31]

5. Secondary Outcome: Overall Survival (OR)
Description: It is defined as the time between the start of study treatment to date of death from any cause. If it were impossible to obtain confirmation of the death, survival will be censored with the date of the last Visit that it is satisfied that the patient was alive.
Time Frame: approximately 36 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | TH-302 + Sunitinib
Number analyzed (Participants) | 17
months | 32.32 [25.12 to 39.53]

6. Secondary Outcome: Safety (Adverse Events)
Description: Safety will be assessed according to the reports of adverse events, the frequency of treatment discontinuations due to adverse events, laboratory evaluations or ECG
Time Frame: time between the date of signing the informed consent until 28 days after the last dose of study drug, , an average of 2 years
Measure: Number; unit: events
Arm/Group | TH-302 + Sunitinib
Number analyzed (Participants) | 17
events
  SAE | 3
  Deaths (all causes) | 3
  Deaths (SAE related) | 1
  AE | 17
  treatment discontinuation due to toxicity | 4

7. Secondary Outcome: Biomarkers in Serum and Tumor Tissue
Description: Assess the predictive/prognostic value of the analysed biomarkers in plasm and tumour.
Time Frame: approximately 36 months
Population: we obtained samples from 13 patients for Cg A and 10 patients for Enolase 1
Measure: Median (Full Range); unit: ng/ml
Arm/Group | TH-302 + Sunitinib
Number analyzed (Participants) | 13
ng/ml
  Cg A | 197 [37.2 to 2063.90]
  Enolase 1: number analyzed (Participants) | 10
  Enolase 1 | 15.06 [8.60 to 92.89]

ADVERSE EVENTS:
Time Frame: The security assessment period was between the date of the signed informed consent and up to 28 days after the last dose of study drug, an average of 2 years
Arm/Group | TH-302 + Sunitinib
All-Cause Mortality (participants affected / at risk) | 3/17
Serious Adverse Events (participants affected / at risk) | 3/17
Other Adverse Events (participants affected / at risk) | 17/17
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | TH-302 + Sunitinib (N=17)
Aspartate aminotransferase increased (Blood and lymphatic system disorders) | 1 (1)
Alanine aminotransferase increased subjects affected / exposed (Blood and lymphatic system disorders) | 1 (1)
Fever (General disorders) | 1 (1)
Fatigue (General disorders) | 1 (1)
Biliary duct obstruction (Hepatobiliary disorders) | 1 (1)
Pancreatitis (Endocrine disorders) | 1 (1) — Death related SAE
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | TH-302 + Sunitinib (N=17)
Hypertension (Vascular disorders) | 6 (6)
Vascular disorders - Other, brachial vein thrombosis (Vascular disorders) | 2 (2)
Fatigue (General disorders) | 14 (14)
General disorders and administration site conditions - Other, epigastralgia (General disorders) | 3 (3)
Fever (General disorders) | 3 (3)
Dizziness (General disorders) | 1 (1)
Abdominal pain (General disorders) | 1 (1)
Depression (Psychiatric disorders) | 1 (1)
Vaginal inflammation (Reproductive system and breast disorders) | 2 (2)
Reproductive system and breast disorders - Other, genital dryness (Reproductive system and breast disorders) | 1 (1)
Mucositis oral (Respiratory, thoracic and mediastinal disorders) | 10 (10)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Respiratory, thoracic and mediastinal disorders - thoracic pain (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Neutrophil count decreased (Blood and lymphatic system disorders) | 9 (9)
Platelet count decreased (Blood and lymphatic system disorders) | 5 (5)
Alanine aminotransferase increased (Blood and lymphatic system disorders) | 3 (3)
Blood bilirubin increased (Blood and lymphatic system disorders) | 2 (2)
Anemia (Blood and lymphatic system disorders) | 2 (2)
White blood cell decreased (Blood and lymphatic system disorders) | 1 (1)
Hypocalcemia (Blood and lymphatic system disorders) | 1 (1)
Bilirrubin increased (Blood and lymphatic system disorders) | 1 (1)
Aspartate aminotransferase increased (Blood and lymphatic system disorders) | 1 (1)
Headache (Nervous system disorders) | 4 (4)
Myalgia (Nervous system disorders) | 2 (2)
Dysesthesia (Nervous system disorders) | 2 (2)
Peripheral motor neuropathy (Nervous system disorders) | 1 (1)
Paresthesia (Nervous system disorders) | 1 (1)
Conjunctivitis (Eye disorders) | 2 (2)
Diarrhea (Gastrointestinal disorders) | 9 (9)
Dyspepsia (Gastrointestinal disorders) | 3 (3)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 2 (2)
Dysphagia (Gastrointestinal disorders) | 2 (2)
Rectal hemorrhage (Gastrointestinal disorders) | 1 (1)
Hemorrhoids (Gastrointestinal disorders) | 1 (1)
Gastrointestinal disorders - Other, specify: aerophagia (Gastrointestinal disorders) | 1 (1)
Gastrointestinal disorders - Other, specify: acute gastroenteritis (Gastrointestinal disorders) | 1 (1)
Gastrointestinal disorders - Other, glossitis (Gastrointestinal disorders) | 1 (1)
Gastrointestinal disorders - Other, Gingivitis (Gastrointestinal disorders) | 1 (1)
Esophagitis (Gastrointestinal disorders) | 1 (1)
Anal ulcer (Gastrointestinal disorders) | 1 (1)
Anal pain (Gastrointestinal disorders) | 1 (1)
Hematuria (Renal and urinary disorders) | 1 (1)
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 5 (5)
Rash acneiform (Skin and subcutaneous tissue disorders) | 4 (4)
Skin hypopigmentation (Skin and subcutaneous tissue disorders) | 2 (2)
Skin and subcutaneous tissue disorders - Other, Erythema (Skin and subcutaneous tissue disorders) | 2 (2)
Skin induration (Skin and subcutaneous tissue disorders) | 1 (1)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 1 (1)
Skin and subcutaneous tissue disorders - Other, specify: Unspecified Onycopathy (Skin and subcutaneous tissue disorders) | 1 (1)
Skin and subcutaneous tissue disorders - Other, specify: Psoriasis (Skin and subcutaneous tissue disorders) | 1 (1)
Skin and subcutaneous tissue disorders - Other, Inguinal cutaneous toxicity (Skin and subcutaneous tissue disorders) | 1 (1)
Skin and subcutaneous tissue disorders - Other, facial rash (Skin and subcutaneous tissue disorders) | 1 (1)
Skin and subcutaneous tissue disorders - Other, eczematous facial rash (Skin and subcutaneous tissue disorders) | 1 (1)
Erythroderma (Skin and subcutaneous tissue disorders) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 7 (7)
Dysgeusia (Metabolism and nutrition disorders) | 6 (6)
Nausea (Metabolism and nutrition disorders) | 5 (5)
Vomiting (Metabolism and nutrition disorders) | 4 (4)
Pancreatitis (Endocrine disorders) | 1 (1)
Constipation (Infections and infestations) | 2 (2)
Pharyngitis (Infections and infestations) | 1 (1)
Nail infection (Infections and infestations) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor commits to the timely dissemination of the results through scientific conferences and publications which will be responsible for the scientific coordinator and the translational study coordinator. The study coordinator reserves the option to choose your position in the different publications and reports that could be carried out of the study. The coordinator of the study will have a secure position within the authors. The rest of IPs will be assigned according to order of recruitment

DOCUMENTS (2):
  • Study Protocol (2016-11-23): https://cdn.clinicaltrials.gov/large-docs/62/NCT02402062/Prot_000.pdf
  • Statistical Analysis Plan (2018-11-12): https://cdn.clinicaltrials.gov/large-docs/62/NCT02402062/SAP_001.pdf